CLINICAL TRIAL: NCT03335605
Title: Improving the Diagnosis of Common Variable Immune Deficiency by Analysis of Innate and Adaptive Signaling Pathways
Brief Title: Improving the Diagnosis of Common Variable Immune Deficiency
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Jeffrey Modell Foundation (Unknown)
Responsible Party: Principal Investigator, Manish J. Butte, MD PhD, Associate Professor and Chief, University of California, Los Angeles
Other Study IDs: UCLA-IMMUNOLOGY-16-001950; NCT02680652 (obsolete NCT alias)
Record Dates: First submitted 2017-10-27; First posted 2017-11-08 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: CVI - Common Variable Immunodeficiency
Keywords: primary immunodeficiency
MeSH Terms: conditions — Common Variable Immunodeficiency; Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — < 5 mL of whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Antibody deficiency (CVID): Subjects with antibody deficiency (CVID)
- Healthy controls: Age and gender-matched control subjects

SUMMARY:
This is an observational, case-control study with a single blood draw among two cohorts, patients with antibody deficiency (e.g., CVID) and healthy controls. Samples will be analyzed by mass cytometry (CyTOF) to examine the major signaling pathways of all circulating innate and adaptive immune cell types, as well as whole exome sequencing. The goal is to improve our general understanding of the human immune response to infections and the diagnosis of CVID.

DETAILED DESCRIPTION:
An increased susceptibility to bacterial and viral infections is the hallmark primary immunodeficiencies (PIDs). The most common PIDs requiring treatment with Ig replacement (SCIg or IVIg) is Common Variable Immune Deficiency (CVID), which is diagnosed by the presence of hypogammaglobulinemia plus defective responses to vaccine antigens. Prior to diagnosis, CVID patients often develop autoimmunity that requires immunosuppression or cancers that require chemotherapy. Unfortunately, difficulties arise in making the diagnosis of CVID in adults treated with immunosuppressive drugs, steroids, or chemotherapy, preventing the timely use of Ig replacement therapies in these patients. Furthermore, CVID is difficult to diagnose in young children. Exome sequencing and other genetic methods have thus far failed to identify clear monogenic causes for CVID. At the same time, patients with derangements of signaling pathways including STAT1, STAT3, NFKB, PI3K, and others, have clinical antibody deficiency, suggesting that by examining the signaling pathways, the investigators could find signs of CVID. The Investigators propose to use a broad, new screen to study the functional defects of human immune responses in CVID. Using time-of-flight mass cytometry (CyTOF) and phospho-specific antibodies, the investigators will simultaneously examine the major signaling pathways of all circulating innate and adaptive immune cell types at once to identify abnormal phosphorylation of signaling molecules in response to a variety of canonical stimuli. This method is innovative because it identifies signaling defects in the immune response while being insensitive to chemotherapy or immunosuppression, because the signaling responses examined are biologically upstream of immunosuppressed targets. Our approach generates a new "signaling fingerprint" for facilitating the diagnosis of CVID. Our proposal is also impactful, because knowledge gained about functional defects in CVID, when combined with whole exome sequencing, will improve the general understanding of the human immune response to infections.

There are two major aims: 1) studying healthy control subjects across a variety of ages as comparisons to CVID patients, and furthermore to generate new information about how immune signaling responses change with age, which is currently unknown; and 2) studying CVID patients to identify the consistent aberrant signaling responses that will allow the acceleration of diagnosis and treatment.

Design of study: The investigators propose an observational, case-control study with a single blood draw among two cohorts, patients with antibody deficiency (CVID) and healthy controls. Methods: Fifty (50) CVID patients (adult and children) will be consented in the Immunology Clinic at UCLA. Healthy, age- and gender-matched controls will be sought at the same time (100). There will be one blood draw of < 5 mL of blood to be analyzed immediately by phospho-CyTOF at UCLA. Genomic DNA will be prepared from samples and sequences analyzed.

This screen examines phosphorylation of all circulating immune cell types at once (CD4 and CD8 T cells, B cells, NK cells, monocytes, macrophages, neutrophils, eosinophils, and DCs). Whole blood from subjects and from controls will be aliquotted into portions, and each portion will be stimulated with either cytokines, TLR agonists, anti-TCR or anti-BCR antibodies, PMA, or left unstimulated. Treated cells will be surface stained, fixed, permeabilized, and stained intracellularly for 12 signaling phospho-proteins, then analyzed by CyTOF, which enables measurement of over 50 parameters simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of antibody deficiency (CVID)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of CVID and Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Differences in Immune Cells in CVID and healthy controls | 2 years
  Whole blood from subjects and from controls will be aliquotted into portions, and each portion will be stimulated with either cytokines, TLR agonists, anti-TCR or anti-BCR antibodies, PMA, or left unstimulated. Treated cells will be surface stained, fixed, permeabilized, and stained intracellularly for 12 signaling phospho-proteins, then analyzed by CyTOF, which enables measurement of over 50 parameters simultaneously across all circulating immune cell types (CD4 and CD8 T cells, B cells, NK cells, monocytes, macrophages, neutrophils, eosinophils, and DCs). All responses across all cells for all stimuli will be aggregated by principal components analysis to a single metric that will be compared between subjects with antibody deficiency and controls.

CONTACTS AND LOCATIONS:
Overall Officials: Manish J Butte, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi J, Fernandez R, Maecker HT, Butte MJ. Systems approach to uncover signaling networks in primary immunodeficiency diseases. J Allergy Clin Immunol. 2017 Sep;140(3):881-884.e8. doi: 10.1016/j.jaci.2017.03.025. Epub 2017 Apr 13. PMID 28412396